CLINICAL TRIAL: NCT07249203
Title: Effects of Resistance Training Applied With a Velocity-Based Approach on Selected Motor Skills
Brief Title: Velocity-Based Resistance Training and Motor Skills in University Athletes
Acronym: VBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGU-2024-01-144-VBT-1
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Resistance Training; Motor Performance; Athletic Performance; Velocity-based Training
Keywords: Velocity-based training, Speed, Agility, Maximal strength, Performance

STUDY DESIGN:
Intervention Model Description: The study employed a parallel-group, randomized design. Participants were randomly assigned to either a percentage-based training (PBT) group or a velocity-based training (VBT) group. Both groups performed resistance training programs for 8 weeks, focusing on lower-body and upper-body exercises. The VBT group trained according to movement velocity feedback, while the PBT group followed loads based on fixed percentages of one-repetition maximum (1RM). Pre- and post-tests were conducted to evaluate changes in motor performance variables such as jump height, sprint time, and maximal strength.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percentage-Based Training (PBT) Group (Experimental): Participants in this group performed a resistance training program based on fixed percentages of their one-repetition maximum (1RM). The training load was adjusted weekly according to percentage-based progression over 8 weeks.
  Interventions: Behavioral: Percentage-Based Training (PBT)
- Velocity-Based Training (VBT) Group (Experimental): Participants in this group performed the same resistance training exercises as the PBT group, but the training load and volume were adjusted according to movement velocity feedback using a linear position transducer. The intervention lasted for 8 weeks.
  Interventions: Behavioral: Velocity-Based Training (VBT)

INTERVENTIONS:
Behavioral: Percentage-Based Training (PBT) — The percentage-based training (PBT) group performed the same resistance exercises as the VBT group for 8 weeks, three sessions per week. Training loads were prescribed according to a fixed percentage of each participant's one-repetition maximum (1RM). Exercises included squats, lunges, and other lower-body movements aimed at improving strength and power.
  Arms: Percentage-Based Training (PBT) Group
Behavioral: Velocity-Based Training (VBT) — The velocity-based training (VBT) group performed lower-body resistance exercises for 8 weeks, three sessions per week. Training loads were adjusted based on real-time barbell velocity feedback measured with a linear encoder. Exercises included squats, lunges, and other multi-joint movements. Each session focused on maintaining optimal movement speed for power development.
  Arms: Velocity-Based Training (VBT) Group

SUMMARY:
This study investigated the effects of resistance training applied with a velocity-based approach on selected motor skills in university-level athletes. Participants were randomly assigned to two groups: a velocity-based training (VBT) group and a percentage-based training (PBT) group. Both groups performed lower-body resistance exercises over an 8-week period, three times per week. Pre- and post-training assessments were conducted for countermovement jump (CMJ), sprint (20 m and 40 m), agility (505 test), and one-repetition maximum (1RM) squat performance. The aim of this study was to compare the effects of VBT and PBT on jump, sprint, agility, and strength performance. It was hypothesized that the VBT group would show greater improvements in motor skills compared to the PBT group.

DETAILED DESCRIPTION:
This randomized, parallel-group, interventional trial was designed to examine the effects of resistance training performed using a velocity-based approach on selected motor skills among trained university athletes.

A total of 20 male participants (aged 18-30 years) were randomly assigned into two groups:

Velocity-Based Training (VBT) group: performed squats, lunges, and similar lower-body exercises using individualized movement velocity feedback obtained from a linear encoder.

Percentage-Based Training (PBT) group: performed the same exercises based on traditional fixed-load percentages of one-repetition maximum (1RM).

Both training programs lasted 8 weeks and included three sessions per week. Pre- and post-tests included measurements of countermovement jump (CMJ) height and power, sprint times (20 m and 40 m), agility (505 test), and maximal squat strength (1RM).

The study was approved by the Istanbul Gelişim University Rectorate Ethics Committee (Approval No: 2024-01-144, Date: 12.01.2024) and conducted in accordance with the Declaration of Helsinki. All participants provided written informed consent prior to participation.

The primary outcome of interest was the change in CMJ performance. Secondary outcomes included sprint, agility, and 1RM strength improvements.

The results are expected to contribute to the understanding of how velocity-based resistance training affects neuromuscular adaptations and physical performance in athletes compared to traditional percentage-based training methods.

ELIGIBILITY:
Inclusion Criteria:

* Male university athletes aged 18-35 years
* Regular participation in resistance training for at least 1 year
* Free from any musculoskeletal injuries during the last 6 months
* Willing to participate in all training sessions and testing procedures

Exclusion Criteria:

* Current or recent musculoskeletal, neurological, or cardiovascular disorders
* Missed more than two training sessions during the study period
* Use of performance-enhancing drugs or supplements during the study
* Any medical condition that prevents participation in resistance training

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Height | 8 weeks (baseline to post-test)
  Countermovement jump height will be measured using a force platform. Jump height (cm) will be calculated from flight time.

SECONDARY OUTCOMES:
20 m Sprint Time | 8 weeks
  Sprint speed will be measured using a 20-meter sprint test with electronic timing gates.
40 m Sprint Time | 8 weeks
  Sprint performance will be measured using a 40-meter sprint test with electronic timing gates.
505 Agility Test Time | 8 weeks
  Change of direction ability will be assessed using the 505 agility test.
1RM Back Squat Strength | 8 weeks
  Maximal lower-body strength will be assessed using the one-repetition maximum (1RM) back squat test.
CMJ Peak Force | 8 weeks
  Peak force (N) during countermovement jump will be measured using a force platform.
CMJ Peak Power | 8 weeks
  Peak power (W) will be calculated using data obtained from the force platform and linear encoder.
CMJ Peak Velocity | 8 weeks
  Peak velocity (m/s) during countermovement jump will be measured using a linear encoder.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar GÜR, PhD, Principal Investigator — Istanbul Gelişim University, Faculty of Sports Sciences
Locations (1):
- Istanbul Gelişim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Summary data may be available from the corresponding author upon reasonable request.

REFERENCES:
- See also: Istanbul Gelişim University official website — https://gelisim.edu.tr/